CLINICAL TRIAL: NCT03629132
Title: Platelet-rich Plasma(PRP) Prevents Recurrence of Intrauterine Adhesions
Brief Title: PRP Prevents Recurrence of Intrauterine Adhesions
Acronym: RPR-IUAs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RPR-IUAs
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia | interventions — Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP (Experimental): Platelet-rich plasma
  Interventions: Procedure: Platelet-rich plasma
- Gel (Sham Comparator): Self-crosslinking sodium hyaluronate gel
  Interventions: Procedure: gel

INTERVENTIONS:
Procedure: Platelet-rich plasma — Platelet-rich plasma intrauterine injection
  Arms: PRP
Procedure: gel — Self-crosslinking sodium hyaluronate gel intrauterine injection
  Arms: Gel

SUMMARY:
Effect of platelet-rich plasma (PRP) on uterine scar fibrosis, endometrial receptivity and pregnancy outcome in patients with severe intrauterine adhesions

DETAILED DESCRIPTION:
1. Inclusion criteria: patients with intrauterine adhesions (AFS score >9 points); age 21 to 40 years old, with fertility requirements.
2. Study design:prospective, randomized controlled cohort study, patients with intrauterine adhesions were randomized into two groups, the control group and the intervention group (intraoperative and postoperative 1 week postoperative PRP). The surgical procedures and postoperative medication regimens were the same.
3. Compare the biochemical pregnancy rate, clinical pregnancy rate, abortion rate and live birth rate after hysteroscopic resection in PRP group and control group, and explore the effect of PRP on pregnancy outcome after intrauterine adhesion.

ELIGIBILITY:
Inclusion Criteria:Patients with intrauterine adhesions (AFS score >9 points); age 21 to 40 years old, with fertility requirements -

Exclusion Criteria:Endometrial tuberculosis, endometrial polyps, uterine submucosal fibroids, endometrial hyperplasia, endometrial malignant lesions, premature ovarian failure, chromosomal abnormalities

-

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
AFS score | 1 year
  AFS score

IPD SHARING:
Plan to Share IPD: No